CLINICAL TRIAL: NCT00625534
Title: Chronic Significant Pain and Functional Outcome After Laparoscopic Versus Open Groin Hernia Mesh Repair: Design of a Randomized Controlled Clinical Trial
Brief Title: Functional Outcome After Groin Hernia Mesh Repair: Open Versus Laparoscopy
Acronym: GENINGHERNIA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Ihsan INAN M.D. Chef de Clinique, Visceral Surgery Division, Department of Surgery, Geneva University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-122
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2008-04

CONDITIONS: Inguinal Hernia; Laparoscopic Surgery; Pain; Sexual Dysfunction, Physiological
Keywords: Hernia; Laparoscopy; Pain; Sexual; Quality
MeSH Terms: conditions — Hernia, Inguinal; Pain; Sexual Dysfunction, Physiological; Hernia; Coitus | interventions — tetraethylpyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Laparoscopic repair
  Interventions: Procedure: Laparoscopic totally extraperitoneal inguinal hernia repair
- 2 (Active Comparator): Open tension free inguinal hernia mesh repair
  Interventions: Procedure: Open tension free inguinal hernia mesh repair

INTERVENTIONS:
Procedure: Laparoscopic totally extraperitoneal inguinal hernia repair — 3 trocars procedure. Blunt camera dissection without use of balloon dissector. Anatomical, preformed, polyester mesh passed around spermatic cord structures. No fixation of mesh.
  Other Names: TEP; Laparoscopic hernia repair
  Arms: 1
Procedure: Open tension free inguinal hernia mesh repair — Classical Lichtenstein repair. Polyester flat 14x8cm mesh
  Other Names: Lichtenstein repair
  Arms: 2

SUMMARY:
Background: Large acceptance of mesh reinforcement techniques in groin hernia repair lowered recurrence rates for all techniques. Recurrence rate alone is not the main quality criterion for hernia repair anymore. Chronic significant post operative pain is a common, clinically relevant, poorly understood and poorly studied entity which is 3 to 5 times more common than hernia recurrence. As a subgroup to chronic significant post operative pain or as a separate entity, sexual dysfunction due to ejaculatory and genital pain after inguinal hernia repair may happen in approximately 2.5% of patients. Patient's preoperative psychological profile as well as pain exposure history is showed to be important in the development of chronic significant post operative pain. The objective of this study is to analyse chronic significant post operative pain and the functional outcome status of patients after laparoscopic repair compared to open repair.

Methods: A randomized controlled non-blinded clinical trial is designed to compare open inguinal hernia mesh repair with laparoscopic totally extraperitoneal repair on chronic significant post operative pain, pain related sexual function disorders, complications, health related quality of life outcomes, recurrence rates, and cost. Volunteers will be recruited in Geneva University Hospital, department of surgery, visceral surgery unit. Eligibility criteria is male patient aged over 21 years, with reducible inguinal unilateral or bilateral primary hernia who are candidates for elective surgery and medically fit for general anesthesia.130 patients will be enrolled for each group to achieve an α-Level of 0.05 and a power of 80%. Follow-up will take place at 10th, 30th days as well as 3 12 and 24 post operative months by questionnaires and by clinical exam by independent expert. An overall cost-analysis will be realized. Patient enrollment in the study will start in April 2008 and estimated to end in may 2009.

DETAILED DESCRIPTION:
Hernia repair is the most frequent elective operation performed in general surgery. Chronic pain or persistent neuralgia has been recognized as a complication after inguinal hernia repair but was reported in the 1980s as a rare and infrequent condition. Studies from the mid 1990s have reported a higher frequency, with up to 50% of patients reporting pain after hernia repair more than 1 year after surgery. Chronic pain after hernia repair can be disabling, with considerable impact on quality of life. The natural history of postoperative pain, including its prevalence, etiology, duration, associated disability and it's social and economical impact remain undefined.

The Cooperative Hernia Study (1996) assessing postoperative pain in a prospective trial including 315 open non-mesh repair patients with 2 years follow-up found at 1 year, 62.9% of groin or inguinal pain and 11.9% of patients had moderate to severe pain; 53.6% had pain and 10.6% of patients continued to report moderate to severe pain 2 years postoperatively.

In a prospective consecutive case series study of 500 consecutive operations in 466 unselected adult patients for open groin hernia repair in Denmark (1994-1996), 1 year after surgery, 19% of patients had some degree of pain, 6% had moderate or severe pain. Pain restricted daily function 6% of patients.

A cross-sectional cohort study based on the Danish Hernia Database (1998) to determine the incidence of groin pain 1 year after inguinal hernia repair and to assess the influence of chronic groin pain on function, detected 28.7% of pain in the groin area and 11.0% of the patients reported that pain was interfering with work or leisure activity. There were no difference in the incidence of pain with regard to the different types of hernia, the different types of surgical repairs, or the different types of anesthesia.

A questionnaire survey of a historical cohort of 351 patients who underwent inguinal hernia surgery in Aberdeen - Scotland (1995-1997) reported 30% chronic pain. Character of this pain was predominantly neuropathic.

Definition of chronic pain The definition of "chronic pain" by the International Association of the Study of Pain is "pain lasting for 3 months or more". There is no consensus on neither in the definition, nor the severity grades of CSPOP in the literature. In the Cooperative Hernia Study, Cunningham et al. clearly described mild, moderate, and severe pain. Mild pain was defined as an occasional pain or discomfort that did not limit activity, with a return to lifestyle before hernia; moderate pain, as pain preventing return to normal preoperative activities (i.e., inability to continue with activities before hernia such as golf, tennis, or other sports, and inability to lift objects without pain, that patients had been lifting before the hernia occurrence); and severe pain, as pain that incapacitated the patient at frequent intervals or interfered with activities of daily living (i.e., a pain constantly present, or intermittently present but so severe as to impair normal activities, such as walking). Other studies defined chronic pain as "that persisting for one year postoperatively". One Dutch study defined pain as pain in the groin or scrotum lasting more than 1 month after surgery. In our study chronic pain is defined as a minimal score > 4 using the quadruple visual analogue scale (VASQ) 3 months after procedure.

Characteristics and etiology of chronic pain Somatic, neuropathic, and visceral chronic pain syndromes are described. Cunningham et al. reported the somatic pain syndrome as the most common type of chronic post hernia pain. The pain is localized to common ligamentous insertion to the pubic tubercle. Somatic pain may be due to the damage to the pubic tubercle during the stapling of mesh prosthesis or from deep muscle layers. Incorporation of the periosteum of the pubic tubercle into the most medial suture during open hernia repair is accused. Neuropathic pain is probably attributable to damage to the ilioinguinal or genitofemoral nerve. Neuropathic pain usually develops in the sensory distribution of an injured nerve. Chronic residual neuralgia occurs as a result of surgical handing of sensory nerves. The nerve trauma can be due to partial or complete division, stretching, contusion, crushing, electrical damage, or sutures compression. Secondary nerve damage can occur due to irritation or compression by an adjacent inflammatory process such as granuloma. Neuropathic pain described as pulling, tugging, tearing, throbbing, stabbing, shooting, numbing, and dull. The onset of neuropathic pain is often delayed, occurring after a latent period of days to weeks. Pain is often aggravated by ambulation, stooping or hyperextension of hip and sexual intercourse; and alleviated by recumbent position and flexion of the hip and thigh. In laparoscopic hernia repair when stapling the mesh, it can penetrate the wall of the inguinal canal entrapping and irritating the sensory nerves. Kinking of the nerves may cause chronic irritation. The third pain syndrome described in the literature is visceral. For example, pain encountered only on ejaculation due to dysfunction of periurethral structures involved in ejaculation. One possible mechanism is the injury to either somatic sacral or sympathetic nerves, resulting in dyssynergia of the ejaculatory effector muscles. It can also be due to stricture in the spermatic duct from the scar tissue or twisting of the cord.

Prognosis of chronic pain Once chronic pain is installed, it does not change without a radical treatment. Cunningham et al. reported a prevalence of mild, moderate, or severe pain of 63% at 1 year postoperatively, which was reduced to 54% after 2 years. Those patients who reported moderate to severe pain at 1 year (12%) continued to report persistent pain at 2 years (11 %).

Risk of developing chronic pain

* Predisposing psychological factors Preoperative psychological state of patient (Depression, dependencies, drug consumption etc.) or history of chronic pain with previous surgery or accident may be a predicting factor.
* Surgical factors Recurrent hernia, preoperative pain and absence of visible bulge before surgery, delayed onset of symptoms after surgery, high pain scores at one week postoperatively and requirement of four or more weeks before returning to work are reported as risk factors for developing of chronic pain.

Impact of surgical technique Several different surgical techniques are studied with each other in the literature and different meta analyses, each with different point of interest, gives different lectures of the reality. Despite the fact that there is no consensus in the literature, surgical technique is clearly one of the key parameters. The overall frequency of chronic pain is higher in studies with specific measurements, where pain is the primary outcome of interest.

* OMR vs. non-mesh repair The hypothetical advantage of tension free repair on chronic pain issue is not confirmed. Two retrospective cohort studies coming from the tenors of open mesh repair, reported less chronic pain with mesh repair. This advantage of mesh repair on pain scores versus conventional no-mesh repairs is not confirmed by randomized controlled trials.
* LR vs. OMR The only study comparing laparoscopic totally extraperitoneal (TEP) repair (Polypropylene mesh without fixation) with classic OMR (Lichtenstein) comes from Kumar et al. They find overall 30% of "chronic pain and discomfort" (22,5% for LR, 38,3% for OMR) after a mean of 21 months post hernia repair. Medical Research Council trial reported a significantly higher incidence of chronic pain after open repair than after laparoscopic repair (37 % versus 29 %) at 1 year. This trial, however, included non-mesh repairs in the open group and transabdominal preperitoneal (TAP) and TEP repairs in the laparoscopic group. In a meta-analysis of randomized controlled trials of laparoscopic and open prosthetic mesh repair of groin hernia, EU Trialists found that chronic pain is less likely to occur after laparoscopic repair than after open repair.
* TEP or TAP? The TAP repair is historically the technique of choice in the north america. Most of the literature compares TAP to another technique. In this technique, flat, heavy weighted polypropylene meshes were used and fixed with staplers or tackers. Peritoneal tears were also closed with the same technique. Higher rates of chronic pain were reported after TAP repair versus TEP repair. Nerve entrapment during these several stapling procedures was probably the main reason. TAP is also strongly associated to "rare but serious vascular and visceral complications". The Medical Research Council trial reported that all serious complications occurred in patients undergoing the TAP approach. Most of the postoperative complications as sepsis on bowel fistula with mesh, mechanical ileus on adherences or port site hernias are seen in TAP repair. In our practice TEP repair is the technique of choice. Dissection is realized without the use of balloon dissector, an anatomic, preformed anatomic polyester mesh implanted without fixation by stapling, tacking or suture.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Diagnosis of primary, unilateral or bilateral, reducible groin hernias
* Medically fit for general anesthesia
* Comprehension and use of French language
* Installed in the geographical region without foreseeable move for two years

Exclusion Criteria:

* Female gender, recurrent hernia
* Ongoing chronic pain syndrome, other than hernia origin
* Coagulation disorders, prophylactic or therapeutic anticoagulation, un able to stop platelet antiaggregation therapy 10 days before surgery
* Previous pelvic surgical procedures contraindicating laparoscopic technique
* American Society of Anesthesiology Class 4 and 5 patients
* Emergency surgery, peritonitis, bowel obstruction, strangulation, perforation
* Mentally ill patients
* Presence of local or systemic infection
* Life expectancy < 2 years
* Any cognitive impairment (Psychiatric disorder, Alzheimer's disease etc.)

Ages: 21 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2008-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Chronic significant post operative pain | preoperative, 10, 30, 90, 365 and 730 postoperative days

SECONDARY OUTCOMES:
Pain related sexual function disorders | preoperative, 10, 30, 90, 365 and 730 postoperative days
Health related quality of life | preoperative, 10, 30, 90, 365 and 730 postoperative days
Neuroticism | preoperative, 10, 30, 90, 365 and 730 postoperative days
Postoperative surgical and medical complications | preoperative, 10, 30, 90, 365 and 730 postoperative days
Recurrence rate | 730th postoperative day
Overall cost analysis | 730th postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Morel, Prof., Study Chair — Geneva University Hospital, Departement of Surgery, Visceral Surgery Division; Ihsan INAN, M.D., Study Director — Geneva University Hospital, Departement of Surgery, Visceral Surgery Division
Locations (1):
- Geneva University Hospital, Department of Surgery, Visceral Surgery Division, Geneva, Switzerland